CLINICAL TRIAL: NCT04158362
Title: Open-label, Randomized, Multicenter, Phase III Study, Comparing Standard Chemotherapy to Standard Combination of Endocrine Therapy With Abemaciclib as Initial Metastatic Treatment Among Patients With Visceral Metastasis of ER+ HER2-breast Cancer, High Burden Disease
Brief Title: Endocrine Therapy With Abemaciclib or Chemotherapy as Initial Metastatic Treatment in ER+/HER2- Breast Cancer
Acronym: AMBRE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/1901; 2019-000260-14 (EudraCT Number)
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer Metastatic
Keywords: Abemaciclib; Breast Cancer; High Burden Disease; Visceral Metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — Paclitaxel; Capecitabine; Letrozole; Anastrozole; abemaciclib

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, multicenter, phase III study, comparing standard chemotherapy to standard combination of endocrine therapy with abemaciclib as initial metastatic treatment among patients with visceral metastasis of ER+ HER2- breast cancer, high burden disease.
  Duration of one cycle of either treatment : 3 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Chemotherapy regimen (Experimental): * Paclitaxel: administrated at the dose of 80 mg/m² as a 1-hour intravenous infusion every week (i.e., D1, D8 and D15) of a 3-week cycle.
  OR
  * Capecitabine: given orally at a dose of 2000 to 2500 mg/m² daily for 14 days followed by a 7-day rest period every 3 weeks.
  Interventions: Drug: Paclitaxel injection; Drug: Capecitabine tablets
- Standard Endocrine therapy (ET) regimen + Abemaciclib (Experimental): * Letrozole: continuous orally administration of 2.5 mg/day (1 tablet/day) OR anastrozole continuous orally administration of 1 mg/day (1 tablet/day) in combination with oral abemaciclib 150 mg (BID: twice a day) continuous for patients NSAI naïve or relapsing >1 year after the end of adjuvant ET.
  OR
  * Fulvestrant: 500 mg intramuscular on D1-D15-D29 (loading dose). Then 500 mg every 28 days (maintenance dose) with oral abemaciclib 150 mg BID continuous for patients relapsing on adjuvant or less than one year after completion of adjuvant NSAI.
  For women with a non-menopausal status at inclusion, a concomitant Luteinizing hormone-releasing hormone (LH-RH) agonist will be administered in combination with ET every 28 days. The LH-RH agonist drug to be used will be left to the investigator's choice.
  Interventions: Drug: Letrozole 2.5mg; Drug: Anastrozole 1mg; Drug: Fulvestrant Prefilled Syringe; Drug: Abemaciclib

INTERVENTIONS:
Drug: Paclitaxel injection — Paclitaxel is administrated at the dose of 80 mg/m² as a 1-hour intravenous infusion every week (i.e., D1, D8 and D15) of a 3-week cycle
  Arms: Standard Chemotherapy regimen
Drug: Capecitabine tablets — Capecitabine is given orally at a dose of 2000 to 2500 mg/m² daily for 14 days followed by a 7-day rest period every 3 weeks
  Arms: Standard Chemotherapy regimen
Drug: Letrozole 2.5mg — Letrozole is administered orally at 2.5 mg/day continuous for patients nonsteroidal aromatase inhibitor naïve or relapsing >1 year after the end of adjuvant endocrine therapy.
  Arms: Standard Endocrine therapy (ET) regimen + Abemaciclib
Drug: Anastrozole 1mg — Anastrozole is administered orally at 1 mg/day continous for patients nonsteroidal aromatase inhibitor (NSAI) naïve or relapsing >1 year after the end of adjuvant endocrine therapy.
  Arms: Standard Endocrine therapy (ET) regimen + Abemaciclib
Drug: Fulvestrant Prefilled Syringe — Fulvestrant is administered at the dose of 500 mg intramuscular on D1-D15-D29 (as a loading dose), and then 500 mg every 28 days (as a maintenance dose) for patients relapsing on adjuvant or less than one year after completion of adjuvant NSAI.
  Arms: Standard Endocrine therapy (ET) regimen + Abemaciclib
Drug: Abemaciclib — Oral 150 mg BID continuous
  Other Names: Verzenios®
  Arms: Standard Endocrine therapy (ET) regimen + Abemaciclib

SUMMARY:
AMBRE is a phase III study comparing two standard treatments as initial metastatic treatment in ER+/HER2- breast cancer (BC) patients with visceral metastasis and high burden disease: Chemotherapy and combination of endocrine therapy with abemaciclib.

DETAILED DESCRIPTION:
The primary objective is to compare the efficacy of standard endocrine therapy + abemaciclib combination versus standard chemotherapy based on progression-free survival (PFS), in patients with visceral metastases of ER+/HER2- breast cancer and high tumor burden.

Patients will be randomly assigned to receive either:

* Standard chemotherapy regimen physician's choice either (paclitaxel or capecitabine)
* Standard endocrine therapy regimen physician's choice + abemaciclib (Letrozole or anastrozole for patients nonsteroidal aromatase inhibitor (NSAI) naïve or relapsing >1 year after the end of adjuvant endocrine therapy, and fulvestrant for patients relapsing on adjuvant or less than one year after completion of adjuvant NSAI)

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any study specific procedures.
2. Female age ≥ 18 years.
3. Performance status, Eastern Cooperative Oncology Group (ECOG) 0-2.
4. Histologically confirmed adenocarcinoma of the breast.
5. Metastatic breast cancer, with liver and/or lung and/or pleural and/or peritoneal metastases with high tumor burden (according to RECIST v1.1) defined as either:

   * visceral involvement of one site with more than 3 lesions,
   * visceral involvement of at least 2 sites,
   * symptomatic ascites or pleural effusion, defined as the need for weekly drainage with visceral measurable metastases,
   * visceral involvement and lactate dehydrogenase (LDH) > Normal value.
6. Patient considered candidate for a first line chemotherapy in metastatic setting by their physician (either capecitabine or paclitaxel) and who may receive first-line endocrine therapy combined with abemaciclib according to the marketed authorization.
7. ER-positive by immunohistochemistry (IHC) (>10%) on primary or metastatic disease.
8. HER2-negative by IHC (score 0 or 1+) and/or Fish/Cish negative.
9. Non-menopausal women will receive LH-RH agonists before starting the endocrine therapy and every 28 days thereafter. It is recommended that LH-RH agonist therapy be started approximately 28 days before the start of hormone therapy.
10. Adequate renal, hepatic, and hematopoietic functions as defined by the following criteria:

    * Absolute Neutrophil Count (ANC) ≥1,500/mm³ or ≥1.5 x 10⁹/L
    * Platelets ≥100,000/mm³ or ≥100 x 10⁹/L
    * Hemoglobin ≥8 g/dL (patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion).
    * Serum Aspartate Transaminase (AST) and serum Alanine Aminotransferase Transaminase (ALT) ≤3 x upper limit of normal (ULN) (<5 ULN if liver metastasis)
    * Total serum bilirubin ≤1.5 x ULN (patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted)
    * Serum creatinine ≤1.5 x ULN or estimated creatinine clearance >60 mL/min as calculated using the standard method for the institution.
11. Women of childbearing potential agreeing to use highly effective contraception during treatment and for 3 weeks following the last dose of abemaciclib or for 6 months following the last dose of capecitabine or paclitaxel or for 2 years following the last dose of fulvestrant.
12. Women of childbearing potential must have a negative serum pregnancy test within 7 days and/or urine pregnancy test 48 hours prior to the administration of any study treatment.
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
14. Health insurance coverage.

Exclusion Criteria:

1. Bone lesion only or non-measurable lesion (RECIST V1.1).
2. Patients with all target lesions in a previously irradiated region, except if clear progression has been observed prior to study in at least one of them.
3. Spinal cord compression and/or symptomatic or progressive brain metastases (Brain metastasis are not acceptable unless asymptomatic or treated and stable off steroids for at least 30 days prior to start of study drug).
4. Patient with visceral crisis as defined in the 4th ESO-ESMO International Consensus Guidelines (severe organ dysfunction as assessed by signs and symptoms, laboratory studies and rapid progression of disease).
5. Patient has received one line of chemotherapy for metastatic disease.
6. Patient has received endocrine therapy for metastatic disease.
7. Inability to swallow orally administered medication.
8. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
9. Major problem with intestinal absorption.
10. Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix or the breast, and adequately treated basal cell or squamous cell carcinoma of the skin.
11. Patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
12. Patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
13. Patient has any serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30 mL/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
14. Any drug or plant derivative that may interact with abemaciclib.
15. Episode of pulmonary thromboembolism (PTE) in the last six months. Patients with deep vein thrombosis previously treated with a low-molecular-weight heparin for more than two months prior enrolment in the study will be eligible.
16. Patients with previously documented total/partial dihydropyrimidine dehydrogenase (DPD) deficiency or with DPD deficiency identified at baseline visit (plasma uracil concentration ≥16 ng/mL). These patients will be not eligible for chemotherapy by capecitabine.
17. Pregnant or breast feeding women.
18. Patients enrolled in another therapeutic study within 30 days prior inclusion.
19. Individuals deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the date of the first documented progression (RECIST v1.1) or death from any cause up to 48 months
  PFS will be measured from the date of randomization until the date of event defined as the first documented progression (RECIST v1.1) or death from any cause.

SECONDARY OUTCOMES:
Patients' quality of life by the Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline and every 6 weeks during 24 weeks
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Patients' quality of life by the Quality of Life Questionnaire - Breast cancer module (QLQ-BR23) | At baseline and every 6 weeks during 24 weeks
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms.
Patients' quality of life by the Quality of Life G8 | At baseline
  The G8 questionnaire is a 8-item screening tool developed specifically for older patients (>70 years old) leaving with cancer. This tool, addressed by the clinician, covers multiple domains, focusing on nutritional status, weight loss, body mass index, mobility, neuropsychological problems, medication use, self-rated health status, and age. The score ranges from 17 (not at all impaired) to 0 (heavily impaired).
Objective response rate (ORR) | 24 weeks
  The overall response rate (ORR) will be defined as the proportion of randomized patients who achieve a complete response (CR) or a partial response (PR) at 24 weeks.
Duration of response (DoR) | evey 8 weeks up to 48 months
  The duration of response (DoR) will be defined as the duration between the time of tumor response (CR or PR) until the date of objective progression.
Progression-free-survival 1 (PFS1) | Throughout the study up to 48 months
  PFS1 is defined as the interval between the date of randomization and the date of progression or death from any cause regardless of whether the patient withdraws from randomized study treatment or receives another anti-cancer therapy prior to progression.
Progression-free-survival 2 (PFS2) | Throughout the study up to 48 months
  PFS2 is defined as the time from the date of randomization to the earliest of the progression event subsequent to that used for the primary variable PFS, or date of death (i.e., objective radiological, CA15-3 or symptomatic progression).
PFS1 and PFS2 in prespecified subgroups defined by stratification factors | Throughout the study up to 48 months
  Stratification will be performed according to:
  1. Sensitivity to Endocrine therapy
     * endocrine sensitive = relapse >1 year after ending adjuvant endocrine therapy
     * endocrine resistance = relapse during or within 1 year after ending adjuvant endocrine therapy
     * de novo
  2. Planned chemotherapy (capecitabine versus paclitaxel)
  3. Liver metastasis Yes or No. Block randomization (ratio 1:1) will be stratified by the 12 (3*2*2) above-described groups
Overall survival (OS) | From the date of randomization to the date of death from any cause, assessed up to 48 months
  The overall survival is the length of time from randomization that patients endocrine therapy/abemaciclib improves overall survival compared to chemotherapy.
Incidence of Treatment-Emergent Adverse Events | Throughout study completion, up to 48 months
  The tolerance and safety will be evaluated by toxicity (acute [<6 months after the start of atezolizumab] and late [≥6 months after the start of atezolizumab]), assessed using the NCI CTCAE v5.0.
Maintenance regimens after chemotherapy regimen | 48 months
  Number of maintenance regimens administered after the end of the standard treatment by chemotherapy and in the absence of disease progression.
Circulating tumor cell (CTC) count | At baseline
  To study the predictive and prognostic value of circulating tumor cell count (<5 versus ≥ 5 CTC/7.5mL)
Progression-free survival (PFS) within 24 weeks | From randomization to the date of the last available tumor assessment up to 24 weeks.
  PFS within 24 months will be measured from the date of randomization until the date of event defined as the first documented progression (RECIST v1.1) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique DIERAS, Dr, Principal Investigator — Centre Eugène Marquis, Rennes; Gilles FREYER, Pr, Principal Investigator — Centre Hospitalier Lyon Sud
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.